CLINICAL TRIAL: NCT07052812
Title: Exploring The Metacognitive Beliefs in OCD: A Randomized Controlled Trial of Metacognitive Therapy
Acronym: MCT-OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Responsible Party: Principal Investigator, Saeed Anwar, Doctoral student, Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022035
Record Dates: First submitted 2025-06-29; First posted 2025-07-07 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2024-01

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: Obsessive-Compulsive Disorder, Metacognitive Beliefs, Metacognitive Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Parallel-Group Model Description:** "This randomized controlled trial employed a two-arm parallel design comparing Metacognitive Therapy (MCT) with standard Treatment As Usual (TAU) for OCD. Participants (N=76) were equally allocated to either: (1) MCT - 12 weekly sessions targeting metacognitive beliefs about thoughts, or (2) TAU - routine care including medications and basic counseling with family involvement. Randomization used computer-generated blocks with allocation concealment. Both groups were assessed identically at baseline, post-treatment (week 12), and 6-month follow-up using Y-BOCS as the primary outcome. The parallel structure ensured no treatment crossover. TAU specifically included supportive counseling (not formal CBT) with family participation in care, reflecting real-world clinical practice in the study settings. Independent assessors, blinded to treatment assignment, conducted all evaluations.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCT (Experimental): Arm Description for "MCT" (Experimental Arm):** "Participants receive 12 weekly sessions of manualized Metacognitive Therapy (MCT) for OCD, delivered by trained clinicians. The intervention targets maladaptive metacognitive beliefs (e.g., thought-action fusion) through: (1) Attention Training Technique, (2) Detached Mindfulness exercises, and (3) behavioral experiments to modify compulsions. Treatment progresses through four phases: psychoeducation, challenging perfectionism, addressing intolerance of uncertainty, and relapse prevention. Primary outcome: Yale-Brown Obsessive Compulsive Scale (Y-BOCS)
  Interventions: Behavioral: MCT
- TAU (Active Comparator): Treatment as Usual (TAU) consists of 12-week standard outpatient care for OCD, including:
  * Psychoeducation about OCD symptoms.
  * Supportive counseling (stress management, coping strategies).
  * SSRI medication management (if prescribed).
  * Simplified exposure exercises (without formal ERP protocols).
  * Family involvement in care.
  Interventions: Behavioral: MCT

INTERVENTIONS:
Behavioral: MCT — Metacognitive Therapy (MCT) is a 12-week manualized treatment for OCD targeting maladaptive thought patterns. Clinicians deliver structured sessions including: (1) Attention Training to modify focus, (2) Detached Mindfulness to change responses to intrusive thoughts, and (3) behavioral experiments to reduce compulsions. Treatment progresses through psychoeducation, challenging perfectionism, addressing thought control, and relapse prevention. Primary outcome: Y-BOCS; secondary: MCQ-30 and TFI. Based on the evidence-based myMCT protocol.

SUMMARY:
Exploring The Metacognitive Beliefs in OCD: A Randomized Controlled Trial of Metacognitive Therapy Introduction Obsessive-Compulsive Disorder (OCD) is a mental health condition characterized by intrusive thoughts (obsessions) and repetitive behaviors (compulsions). These symptoms cause significant distress and impair daily functioning. OCD can be difficult to treat, and relapse rates are high even after conventional treatments. This study evaluates whether Metacognitive Therapy (MCT) is more effective than Treatment as Usual (TAU) in reducing OCD symptoms and improving overall well-being. The study explores how MCT, which targets metacognitive beliefs (thoughts about thoughts), can help manage symptoms more effectively than standard treatments.

Study Goal and Research Question

The primary goal of this study is to assess the effectiveness of Metacognitive Therapy (MCT) compared to Treatment as Usual (TAU) for treating Obsessive-Compulsive Disorder (OCD). The key research question is:

Does Metacognitive Therapy (MCT) reduce OCD symptoms more effectively than Treatment as Usual (TAU)? Study Design

This study is a Randomized Controlled Trial (RCT), which means participants are randomly assigned to one of two treatment groups:

Metacognitive Therapy (MCT): Participants in this group receive a 12-session therapy program that focuses on addressing harmful metacognitive beliefs, such as the need to control thoughts and the belief that thoughts can cause harm.

Treatment as Usual (TAU): Participants in this group receive the standard treatment for OCD, which may include Exposure and Response Prevention (ERP) and/or medication.

Who Can Participate? Adults aged 18 and older who have been diagnosed with OCD are eligible to participate in the study. To be eligible, participants must have moderate to severe OCD symptoms, measured by the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). Individuals with severe mental health conditions other than OCD, such as psychosis or substance use disorders, are excluded from participation. Participants must also be able to attend therapy sessions and complete the necessary assessments throughout the study.

How the Study Was Conducted Randomization: Participants were randomly assigned to either the MCT group or the TAU group.

MCT Group: Participants in the MCT group attended 12 therapy sessions, which focused on changing metacognitive beliefs that contribute to OCD symptoms.

TAU Group: Participants in the TAU group received standard treatment for OCD, which may have included a combination of therapy and medications.

Assessments: Participants were assessed at three time points: before treatment (pre-treatment), immediately after treatment (post-treatment), and six months after treatment (follow-up). These assessments measured changes in OCD symptoms, metacognitive beliefs, and overall quality of life.

Study Procedures and Timeline Pre-Treatment Assessment: Participants completed initial assessments to measure their OCD symptoms, metacognitive beliefs, and quality of life.

Therapy Sessions: Participants in both groups attended their respective therapy sessions (12 sessions for MCT, standard sessions for TAU).

Post-Treatment and Follow-Up Assessments: After the therapy ended, participants completed post-treatment assessments. Six months later, they participated in a follow-up assessment to measure the long-term effectiveness of the treatment.

Important Information for Participants Metacognitive Therapy (MCT) is designed to help people change the way they think about their thoughts, addressing beliefs such as the need to control thoughts or the belief that having certain thoughts can cause harm.

Treatment as Usual (TAU) is the standard treatment for OCD, which may include Exposure and Response Prevention (ERP) therapy or medication management.

Participants in this study can withdraw at any time, and their decision will not affect their treatment or relationship with their healthcare provider.

Expected Benefits If MCT is found to be more effective than TAU, it may offer a new, personalized approach to treating OCD, especially for individuals whose symptoms are driven by dysfunctional metacognitive beliefs. Additionally, since MCT targets the underlying thought processes that maintain OCD symptoms, it may provide longer-lasting symptom relief and reduce the likelihood of relapse compared to standard treatments.

Study Impact This study will provide important insights into whether MCT can provide better outcomes for individuals with OCD compared to standard treatments. If MCT is shown to be effective, it could become a valuable treatment option for those who do not respond well to traditional therapies like ERP. Moreover, MCT's focus on addressing metacognitive beliefs may lead to more durable improvements in OCD symptoms.

DETAILED DESCRIPTION:
Introduction:

Obsessive-Compulsive Disorder (OCD) is a chronic, debilitating mental health condition that affects approximately 1-2% of the global population. It is characterized by obsessions, which are intrusive and unwanted thoughts, images, or urges, and compulsions, which are repetitive behaviors or mental acts performed to neutralize or reduce the anxiety caused by the obsessions. These symptoms not only lead to significant personal distress but also impair social, occupational, and academic functioning, severely affecting quality of life.

OCD is considered a complex disorder with a range of symptom severity, from mild and transient symptoms to extreme and persistent disturbances that severely disrupt daily life. The clinical presentation of OCD varies widely, with individuals experiencing different combinations of obsessions and compulsions. For example, some individuals primarily experience contamination fears and engage in cleaning compulsions, while others may have intrusive, violent thoughts associated with compulsions like checking or hoarding. Despite the heterogeneity in symptom presentation, individuals with OCD share a common experience of cognitive intrusiveness, which fuels distress and leads to compulsive behavior aimed at reducing this distress.

While the exact cause of OCD remains unclear, research suggests that the disorder arises from a complex interaction of genetic, neurobiological, and environmental factors. Functional imaging studies have implicated abnormalities in the fronto-striatal circuits, including areas such as the orbital frontal cortex, caudate nucleus, and thalamus, which are involved in cognitive control, impulse inhibition, and habit formation. These abnormalities contribute to dysfunctional cognitive processing, which is thought to lead to the obsessions and compulsions characteristic of OCD.

Standard Treatment Approaches for OCD The most widely recognized treatments for OCD include Cognitive Behavioral Therapy (CBT) and pharmacotherapy, primarily Selective Serotonin Reuptake Inhibitors (SSRIs). Exposure and Response Prevention (ERP), a form of CBT, is considered the gold standard for OCD treatment. ERP involves exposing individuals to feared stimuli or situations (i.e., their obsessions) while preventing them from engaging in the corresponding compulsive behaviors (i.e., the rituals designed to reduce anxiety). This process helps individuals learn that their anxiety decreases naturally over time without the need for compulsions, which ultimately breaks the cycle of obsession and compulsion.

For patients who do not respond to ERP alone, pharmacotherapy-particularly SSRIs, such as fluoxetine, sertraline, and fluvoxamine is often used to enhance symptom relief. Studies have shown that SSRIs can significantly reduce OCD symptoms by increasing serotonin availability in the brain, which helps regulate mood and anxiety levels. However, even with these treatment options, a significant proportion of individuals with OCD continue to experience residual symptoms, and relapse rates remain high, indicating the need for additional or alternative therapeutic approaches.

Despite these advances, treatment outcomes for OCD remain suboptimal for a subset of patients. Approximately 40% of individuals with OCD do not respond adequately to first-line treatments like CBT and SSRIs. Relapse following treatment cessation is also a significant issue, with many individuals experiencing symptom recurrence after achieving initial symptom relief. This suggests that traditional treatments often fail to address underlying cognitive processes that sustain OCD symptoms.

The Role of Metacognitive Beliefs in OCD Recent advancements in cognitive theory have provided insight into the cognitive mechanisms that maintain OCD symptoms. One key area of focus is the role of metacognitive beliefs. Metacognition refers to the cognitive processes we use to think about and monitor our own thoughts, and how we regulate, control, and reflect on them. Metacognitive beliefs are defined as beliefs about one's cognitive processes, such as the perception that certain thoughts are uncontrollable, dangerous, or harmful.

For individuals with OCD, metacognitive beliefs can be a driving force behind obsessive thinking and compulsive behaviors. People with OCD often believe that having a certain thought will result in negative consequences (e.g., "If I think about harming someone, I will act on it") or that they must control their thoughts to avoid harm (e.g., "I must prevent all violent thoughts to keep my family safe"). These types of beliefs not only contribute to the development of OCD but also perpetuate the cycle of obsession and compulsion.

Metacognitive Therapy (MCT), developed by Adrian Wells, focuses on modifying these dysfunctional metacognitive beliefs. The goal of MCT is to help individuals with OCD recognize that their thoughts do not need to be controlled or avoided. Instead, MCT helps individuals develop a more flexible and less reactive relationship with their thoughts, ultimately reducing the need for compulsive behaviors. This approach aligns with the Self-Regulatory Executive Function (S-REF) model, which posits that dysfunctional metacognitive beliefs lead individuals to engage in unhelpful cognitive strategies (e.g., thought suppression, rumination) that maintain OCD symptoms.

Metacognitive Therapy (MCT) as a Treatment for OCD Metacognitive Therapy (MCT) offers an innovative treatment approach for OCD by focusing on the metacognitive processes that sustain obsessive thinking. MCT operates under the assumption that OCD is maintained not only by the content of intrusive thoughts but also by the cognitive strategies individuals use to manage these thoughts, such as thought suppression and rumination. These strategies are often maladaptive and ultimately reinforce the OCD cycle.

MCT aims to challenge and change dysfunctional metacognitive beliefs by helping individuals with OCD:

Recognize and understand their metacognitive beliefs about thoughts (e.g., "I must control my thoughts at all costs").

Learn that thoughts are not inherently dangerous and that attempting to control thoughts often exacerbates anxiety.

Develop alternative coping strategies that reduce the need for compulsions, such as adopting a more flexible relationship with thoughts through techniques like mindfulness and detached observation.

A central component of MCT is helping individuals to accept intrusive thoughts rather than engage in thought control or compulsive behavior. By learning that thoughts are not inherently threatening, individuals can break free from the need to neutralize or avoid certain thoughts. This process is supported by behavioral experiments, in which participants are gradually exposed to feared thoughts or situations while refraining from compulsions.

The current study investigates whether MCT provides superior outcomes compared to TAU, which often includes ERP and pharmacotherapy. We hypothesize that MCT will provide more substantial symptom relief, lasting effects, and improvements in quality of life for individuals with OCD.

The Need for the Current Study Despite the significant advances in OCD treatment, many individuals remain resistant to standard interventions. Relapse after treatment cessation is common, and the long-term effectiveness of treatments like ERP and pharmacotherapy has been questioned in some cases. This underscores the importance of exploring alternative therapeutic approaches that target the underlying cognitive processes involved in OCD.

Metacognitive Therapy offers an innovative approach by addressing the cognitive mechanisms that drive OCD. Given its success in other anxiety disorders, the present study aims to assess the effectiveness of MCT in reducing OCD symptoms compared to the traditional treatment approaches. Specifically, this trial seeks to determine whether MCT leads to greater improvements in symptoms, metacognitive beliefs, and quality of life compared to Treatment as Usual (TAU).

1. Study Design This study is a randomized controlled trial (RCT) designed to evaluate the effectiveness of Metacognitive Therapy (MCT) compared to Treatment as Usual (TAU) for the treatment of Obsessive-Compulsive Disorder (OCD). The study is conducted with two treatment arms: MCT and TAU, with participants randomly assigned to one of the two treatment groups. The RCT design is considered the gold standard for assessing the efficacy of interventions, as it minimizes bias and ensures robust, reliable results.

   The participants are randomly allocated to one of two groups, ensuring equal distribution of baseline characteristics such as OCD severity, age, and gender. The randomization process is conducted using a computer-generated sequence to prevent selection bias and ensure that treatment effects are attributable to the intervention itself, not to external factors.

   Outcome assessors are blinded to participants' treatment allocation to minimize bias in measuring treatment outcomes. However, blinding of participants is not possible because of the nature of the interventions (i.e., participants know whether they are receiving MCT or TAU). This type of single-blind design ensures that outcome measurements are unbiased and strictly dependent on the treatment received.

   Follow-up Schedule

   Assessments occur at three key time points:

   Pre-treatment (baseline): Prior to starting therapy, participants complete a comprehensive assessment of OCD symptoms, metacognitive beliefs, and quality of life.

   Post-treatment (12 weeks): After the completion of 12 weekly therapy sessions, participants are re-assessed to determine changes in OCD symptoms, metacognitive beliefs, and overall quality of life.

   Six-month follow-up: Participants are re-assessed six months after treatment completion to examine the long-term sustainability of treatment effects.

   The follow-up period helps assess whether the benefits of MCT are sustained over time, providing valuable insights into the long-term efficacy of the intervention.
2. Participants Participants were recruited from outpatient mental health clinics specializing in OCD treatment. Informed consent was obtained from all participants prior to their enrollment in the study.

   Eligibility Criteria

   Inclusion Criteria:

   Age: Adults aged 18-65 years. Diagnosis: A confirmed diagnosis of Obsessive-Compulsive Disorder (OCD) according to the DSM-5 criteria.

   Severity: A baseline Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) score of 16 or higher, indicating moderate to severe OCD symptoms.

   Informed Consent: Participants must be able to provide informed consent and fully engage in the therapy and assessment process.

   Exclusion Criteria:

   Severe Comorbid Psychiatric Disorders: Such as psychosis, bipolar disorder, or major depressive disorder that would interfere with participation in the study or require immediate treatment.

   Substance Use Disorders: Current or past substance use disorders or substance abuse that could confound the study's results.

   Cognitive Impairments: Significant cognitive impairments that would prevent the participant from completing self-report measures or engaging fully in therapy.

   Changes in Medication: Participants who have had changes in psychotropic medications within six weeks of study enrollment are excluded, to control for potential confounding effects.

   A total of 76 participants were recruited and randomly assigned to either the MCT group or the TAU group. Randomization was performed using block randomization to ensure balanced group sizes across both treatment arms.
3. Treatment Protocols Metacognitive Therapy (MCT) Group Participants in the MCT group received 12 weekly sessions (each lasting 60 minutes) of Metacognitive Therapy (MCT). The therapy aimed to modify dysfunctional metacognitive beliefs that sustain OCD symptoms, such as the belief that intrusive thoughts are dangerous or must be controlled.

   The MCT treatment protocol was based on the Self-Regulatory Executive Function (S-REF) model, which emphasizes the role of metacognitive beliefs in the regulation of obsessive thinking and compulsive behavior. The therapy protocol included:

   Psychoeducation (Sessions 1-2): Participants were introduced to the concepts of OCD, the role of metacognitive beliefs in maintaining OCD symptoms, and the S-REF model. Psychoeducation aimed to help participants understand the mechanisms of their disorder and how their thoughts influence their anxiety and compulsive behaviors.

   Cognitive Restructuring (Sessions 3-5): Participants identified and challenged harmful metacognitive beliefs, such as the need to control thoughts or the belief that certain thoughts are inherently dangerous. They were taught to reframe these beliefs and develop a more flexible relationship with their thoughts.

   Detached Mindfulness (Sessions 6-8): Mindfulness techniques were introduced to help participants observe their thoughts without engaging in them or trying to suppress them. This approach reduces the emotional impact of intrusive thoughts and decreases the urge to perform compulsions.

   Behavioral Experiments (Sessions 9-12): Participants engaged in behavioral experiments in which they were exposed to feared situations or thoughts but refrained from performing compulsive behaviors. This helped them test the validity of their metacognitive beliefs and learn that their anxiety would decrease naturally over time, without the need for compulsions.

   Treatment as Usual (TAU) Group The TAU group received standard care for OCD, which primarily involved Exposure and Response Prevention (ERP) therapy. ERP is a widely used and evidence-based treatment for OCD, where individuals are gradually exposed to situations or thoughts that trigger anxiety, but they are prevented from performing the corresponding compulsive behaviors.

   Exposure: The primary focus of ERP is exposure to feared stimuli, whether internal (such as intrusive thoughts) or external (such as dirty objects or contamination). Exposure exercises were tailored to each individual's specific OCD symptoms.

   Response Prevention: Participants were encouraged to refrain from engaging in compulsive behaviors during exposure. By doing so, they could learn that their anxiety decreases naturally over time without the need to perform rituals or compulsions.

   In addition to ERP, participants in the TAU group received pharmacotherapy if clinically indicated. This generally involved SSRIs or other medications that can help reduce anxiety and depressive symptoms, which are often co-occurring in OCD patients.
4. Outcome Measures

   Primary Outcome:

   Yale-Brown Obsessive-Compulsive Scale (Y-BOCS): This clinician-administered scale assesses the severity of both obsessive and compulsive symptoms. The total score ranges from 0 (no symptoms) to 40 (severe symptoms). The Y-BOCS is considered the gold standard for measuring OCD severity.

   Secondary Outcomes:

   Metacognitive Beliefs:

   Metacognitions Questionnaire-30 (MCQ-30): This self-report measure assesses beliefs about the uncontrollability of thoughts, the need to control thoughts, and cognitive confidence.

   Obsessional Beliefs Questionnaire-44 (OBQ-44): This tool evaluates obsessive beliefs such as responsibility for harm, thought-action fusion (the belief that thoughts can lead to actions), and the need for thought control.

   Quality of Life:

   World Health Organization Quality of Life (WHOQOL-BREF): This tool assesses overall quality of life across four domains: physical health, psychological well-being, social relationships, and environmental factors. The WHOQOL-BREF is widely used in clinical research to assess the impact of treatment on quality of life.

   Additional Measures:

   Patient Satisfaction: A self-report questionnaire was used to assess satisfaction with the therapy and perceived treatment effectiveness.

   Therapist Adherence: This was monitored through recorded therapy sessions and feedback from the study supervisor to ensure consistency in treatment delivery.
5. Statistical Analysis The data were analyzed using repeated-measures analysis of variance (ANOVA), which compared changes in OCD symptoms, metacognitive beliefs, and quality of life at pre-treatment, post-treatment, and follow-up. The Intention-to-Treat (ITT) approach was used to ensure that all randomized participants were included in the analysis, regardless of treatment adherence. This approach helped preserve the randomization process and minimized biases introduced by dropouts or incomplete data.

Key Statistical Procedures:

Between-Group Comparisons: Analysis of Covariance (ANCOVA) was employed to compare the two treatment groups (MCT vs. TAU) while controlling for baseline differences in OCD severity and other potential covariates, such as comorbid conditions.

Effect Size Calculation: Cohen's d was used to calculate the magnitude of treatment effects. An effect size of 0.8 or greater was considered a large effect size, signifying a substantial treatment effect.

Post-Hoc Analysis: Additional subgroup analyses explored whether baseline factors (e.g., age, gender, baseline OCD severity) influenced treatment outcomes. A total of 76 participants were recruited and randomized into the two treatment groups: MCT (38 participants) and TAU (38 participants). By the end of the study, 73 participants completed the treatment, with 3 participants dropping out due to personal reasons. The groups were balanced in terms of demographic characteristics, including age, gender, and baseline OCD severity as measured by the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). The groups were also similar in terms of comorbid conditions, with 25% of participants in each group having a co-occurring anxiety or mood disorder. The mean age of participants in the MCT group was 34.2 years (SD = 6.3), and 33.8 years (SD = 6.5) in the TAU group. The gender distribution was balanced, with 60% female participants in both groups. The baseline Y-BOCS scores were 29.6 (SD = 6.8) for the MCT group and 30.4 (SD = 7.2) for the TAU group, indicating moderate to severe OCD symptoms at the start of the study.

The Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) was used to measure the primary outcome of OCD symptoms. The MCT group showed a significantly greater reduction in OCD symptoms compared to the TAU group. In the MCT group, the baseline mean Y-BOCS score was 29.6 (SD = 6.8). At post-treatment, the mean Y-BOCS score decreased to 19.2 (SD = 5.3), reflecting a mean reduction of 10.4 points (p < 0.01). At the six-month follow-up, the reduction was sustained, with a mean score of 20.4 (SD = 6.2), resulting in a mean decrease of 9.2 points (p < 0.01), indicating the lasting effect of MCT. In contrast, the TAU group showed a mean reduction of 6.8 points from the pre-treatment baseline (p < 0.05). The baseline mean Y-BOCS score for the TAU group was 30.4 (SD = 7.2), which decreased to 23.6 (SD = 6.7) at post-treatment. At the six-month follow-up, the mean score increased slightly to 26.0 (SD = 7.3), indicating a smaller, less sustained reduction with a mean decrease of 4.5 points (p < 0.05). The between-group comparison showed that the MCT group had significantly greater reductions in OCD symptoms compared to the TAU group, with a larger and more sustained improvement at the six-month follow-up (p < 0.05).

For secondary outcomes, the Metacognitions Questionnaire-30 (MCQ-30) and the Obsessional Beliefs Questionnaire-44 (OBQ-44) were used to measure metacognitive beliefs. The MCT group showed significant improvements in these beliefs. The MCQ-30 baseline score was 76.3 (SD = 13.4) for the MCT group. Post-treatment, the mean score decreased to 62.0 (SD = 11.8), reflecting a mean reduction of 14.3 points (p < 0.01). At the six-month follow-up, the mean score remained low at 64.5 (SD = 12.5), showing that the improvement was maintained. Similarly, the OBQ-44 baseline score was 110.2 (SD = 24.3) for the MCT group. After treatment, the mean score decreased to 97.4 (SD = 20.9), reflecting a mean reduction of 12.8 points (p < 0.01). At follow-up, the score remained at 98.8 (SD = 21.6), indicating continued improvement. In the TAU group, the MCQ-30 baseline score was 77.2 (SD = 15.3), which decreased to 69.4 (SD = 12.6) post-treatment, with a mean reduction of 8.5 points (p < 0.05). However, at follow-up, the mean score increased to 74.1 (SD = 14.2), suggesting some relapse in metacognitive beliefs. For the OBQ-44, the baseline score in the TAU group was 113.5 (SD = 26.1), which decreased to 106.3 (SD = 22.4) post-treatment, reflecting a mean reduction of 7.2 points (p < 0.05). At follow-up, the mean score increased to 110.2 (SD = 23.1), showing partial relapse. Between-group comparisons revealed that the MCT group had significantly greater reductions in both the MCQ-30 and OBQ-44 compared to the TAU group (p < 0.01 for both).

Quality of life was assessed using the World Health Organization Quality of Life (WHOQOL-BREF). The MCT group showed greater improvements across all domains compared to the TAU group. For physical health, the MCT group had a baseline score of 47.2 (SD = 12.3), which increased to 53.7 (SD = 10.1) post-treatment, reflecting a mean improvement of 6.5 points (p < 0.01). At follow-up, the score remained at 54.8 (SD = 11.3). For psychological health, the baseline score was 50.6 (SD = 11.8), and post-treatment, the score improved to 56.4 (SD = 10.2), with a mean improvement of 5.8 points (p < 0.01). At follow-up, the score remained at 55.8 (SD = 10.5). For social relationships, the baseline score was 52.0 (SD = 9.3), and the score improved to 55.2 (SD = 9.1) post-treatment, with a mean improvement of 3.2 points (p < 0.05). At follow-up, the score remained at 54.9 (SD = 9.5). For environmental factors, the baseline score was 51.6 (SD = 10.7), and post-treatment, the score increased to 55.8 (SD = 9.8), reflecting a mean improvement of 4.2 points (p < 0.05). The score remained high at 54.7 (SD = 9.4) at follow-up.

In the TAU group, quality of life improvements were smaller. For physical health, the baseline score was 46.8 (SD = 13.0), which improved to 50.3 (SD = 11.6) post-treatment, reflecting a mean improvement of 3.5 points (p < 0.05). At follow-up, the score decreased to 49.1 (SD = 12.4). For psychological health, the baseline score was 48.5 (SD = 12.5), and post-treatment, the score improved to 52.4 (SD = 10.3), with a mean improvement of 3.9 points (p < 0.05). At follow-up, the score remained at 51.3 (SD = 10.1). For social relationships, the baseline score was 50.1 (SD = 8.7), and the score improved to 52.6 (SD = 9.4) post-treatment, reflecting a mean improvement of 2.5 points (p < 0.05). At follow-up, the score remained at 52.2 (SD = 9.2). For environmental factors, the baseline score was 50.8 (SD = 10.3), and post-treatment, the score improved to 53.1 (SD = 9.8), reflecting a mean improvement of 2.3 points (p < 0.05). However, at follow-up, the score decreased slightly to 51.9 (SD = 10.2).

Between-group comparisons revealed that the MCT group showed significantly greater improvements in physical health, psychological health, and environmental factors (p < 0.01 for physical and psychological health, p < 0.05 for environmental factors), compared to the TAU group. The results of this study provide compelling evidence that Metacognitive Therapy (MCT) is a significantly more effective treatment for Obsessive-Compulsive Disorder (OCD) compared to Treatment as Usual (TAU). Participants in the MCT group demonstrated greater reductions in OCD symptoms, significant improvements in metacognitive beliefs, and sustained benefits in quality of life compared to the TAU group. These findings suggest that targeting the underlying metacognitive processes in OCD, rather than solely focusing on the content of obsessions and compulsions, may offer a more effective and enduring solution to the disorder.

Effectiveness of MCT in Reducing OCD Symptoms The primary outcome of this study was the reduction in OCD symptoms, as measured by the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). The MCT group showed a mean reduction of 10.4 points from baseline to post-treatment, and this improvement was sustained at six-month follow-up with a mean reduction of 9.2 points. These results are highly significant, with p-values well below the threshold for statistical significance (p < 0.01), indicating that the MCT group experienced substantial and lasting symptom relief. In contrast, the TAU group demonstrated a smaller reduction in symptoms, with a mean reduction of 6.8 points at post-treatment, and a smaller improvement of 4.5 points at follow-up, suggesting that the benefits of TAU, which primarily includes Exposure and Response Prevention (ERP) and pharmacotherapy, were more transient.

These findings align with previous research demonstrating that while ERP is the gold standard for OCD treatment, its effects can be limited for some individuals. Studies have found that up to 40% of individuals with OCD fail to achieve full symptom remission with ERP alone. Moreover, relapse rates after ERP treatment are high, with many patients experiencing a return of symptoms over time. In contrast, the sustained reduction in OCD symptoms observed in the MCT group suggests that the modification of metacognitive beliefs may be a crucial factor in preventing relapse and ensuring long-term symptom management. The ability of MCT to address the cognitive processes that maintain OCD-specifically the beliefs about thought control and the need to prevent perceived threats-likely contributes to its superior and enduring effects.

Metacognitive Beliefs and their Role in OCD The secondary outcomes of this study, which focused on changes in metacognitive beliefs, further support the effectiveness of MCT. Participants in the MCT group showed significant reductions in metacognitive beliefs, as measured by the Metacognitions Questionnaire-30 (MCQ-30) and the Obsessional Beliefs Questionnaire-44 (OBQ-44). The mean reduction of 14.3 points on the MCQ-30 and 12.8 points on the OBQ-44 were both highly significant (p < 0.01), and these improvements were sustained at follow-up, indicating that MCT effectively targets the cognitive mechanisms that sustain OCD symptoms.

The reduction in metacognitive beliefs observed in the MCT group suggests that the therapy successfully addresses the underlying thought patterns that maintain OCD. The beliefs that thoughts are dangerous, that intrusive thoughts must be controlled, or that thoughts can lead to harmful outcomes are central to OCD. In this study, MCT helped participants develop a more flexible relationship with their thoughts and reduced the need to engage in compulsions to neutralize these thoughts. This finding is consistent with the Self-Regulatory Executive Function (S-REF) model, which posits that metacognitive beliefs play a key role in the cognitive strategies individuals with OCD use to regulate their thoughts and emotions. By changing these beliefs, MCT reduces the need for thought control and, in turn, decreases the urge to perform compulsive behaviors.

In contrast, the TAU group demonstrated smaller reductions in metacognitive beliefs-8.5 points on the MCQ-30 and 7.2 points on the OBQ-44, with some relapse observed at follow-up. This suggests that Exposure and Response Prevention (ERP), while effective in reducing OCD symptoms, does not fully address the underlying cognitive processes that contribute to the maintenance of the disorder. ERP focuses primarily on confronting the content of intrusive thoughts and preventing compulsive behaviors, but it does not specifically target the beliefs that individuals hold about their thoughts. Therefore, it is not surprising that the TAU group showed smaller and less sustained improvements in metacognitive beliefs.

Quality of Life Improvements The improvements in quality of life observed in the MCT group were also noteworthy. Participants in the MCT group reported significant increases in physical health, psychological health, social relationships, and environmental factors, as measured by the WHOQOL-BREF. These improvements were consistent with the reduction in OCD symptoms, suggesting that as OCD symptoms diminished, participants experienced a broader enhancement in their overall well-being. For example, the mean improvement of 6.5 points in physical health (p < 0.01) and 5.8 points in psychological health (p < 0.01) in the MCT group reflect substantial gains in both physical and emotional well-being. The improvement in social relationships (mean increase of 3.2 points, p < 0.05) and environmental factors (mean increase of 4.2 points, p < 0.05) further underscore the positive impact of MCT on participants' overall quality of life.

These findings are consistent with the literature on OCD treatment, which shows that effective symptom relief is often associated with improvements in quality of life. OCD symptoms-particularly those involving excessive worry, rumination, and compulsive behaviors-can significantly impair social, occupational, and personal functioning. Therefore, it is not surprising that reducing these symptoms leads to improvements in quality of life. However, it is noteworthy that the TAU group also showed improvements in quality of life, although the improvements were smaller compared to the MCT group. The mean improvement in physical health was 3.5 points (p < 0.05), and psychological health showed a mean improvement of 3.9 points (p < 0.05). While these changes are positive, they are less pronounced than those observed in the MCT group, suggesting that the improvements in quality of life may be more limited in the TAU group due to the partial symptom relief provided by ERP alone.

Sustained Treatment Effects and Long-Term Benefits One of the key findings from this study is the sustained nature of the treatment effects in the MCT group. While both the MCT and TAU groups showed improvements in OCD symptoms, the MCT group experienced greater and more lasting improvements at follow-up. This suggests that MCT not only provides short-term relief but also has the potential to offer long-term benefits. In contrast, the TAU group demonstrated some symptom relapse at the six-month follow-up, with OCD symptoms partially returning. This highlights the importance of targeting underlying cognitive processes in OCD treatment and suggests that MCT may be more effective at preventing relapse by addressing the core mechanisms that drive the disorder.

The sustained improvements in the MCT group could be attributed to the focus on changing metacognitive beliefs, which are fundamental to the persistence of OCD symptoms. By helping participants develop a more flexible relationship with their thoughts and reducing their reliance on compulsive behaviors, MCT provides long-term symptom relief that is not simply a temporary reduction in symptoms but rather a lasting change in the cognitive processes that maintain the disorder.

Clinical Implications The findings of this study have important clinical implications for the treatment of OCD. Metacognitive Therapy (MCT) offers a promising alternative or complement to Exposure and Response Prevention (ERP), especially for individuals who do not respond well to traditional therapies or who experience relapse after treatment. MCT targets the cognitive mechanisms that sustain OCD, such as metacognitive beliefs about the uncontrollability of thoughts and the need for thought control, which are not fully addressed by ERP alone.

ELIGIBILITY:
Inclusion Criteria:

* 1. Primary DSM-5 diagnosis of OCD (confirmed by SCID-5) 2. Age 18-65 years 3. Y-BOCS score ≥16 (moderate-to-severe symptoms) 4. Stable medication regimen (no changes in past 6 weeks) 5. Fluent in Urdu or English 6. Willing to attend all sessions and assessments

Exclusion Criteria:

* 1. Current psychotic, bipolar, or severe depressive disorder 2. Active substance use disorder requiring treatment 3. Intellectual disability or cognitive impairment 4. Concurrent psychotherapy for OCD 5. Recent medication changes (past 6 weeks) 6. Completed OCD-specific therapy in past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) total score | Baseline, Week 12 (post-treatment), 6-month follow-up
  The Y-BOCS is a 10-item clinician-rated scale (scores 0-40) measuring OCD symptom severity. Higher scores indicate worse symptoms. Assessed at baseline, post-treatment (week 12), and 6-month follow-up. Primary endpoint is baseline to week 12 change.

SECONDARY OUTCOMES:
Change in Metacognitions Questionnaire-30 (MCQ-30) total score | Baseline, Week 12 (post-treatment), 6-month follow-up
  The MCQ-30 assesses metacognitive beliefs (30 items, scored 30-120). Higher scores indicate more dysfunctional metacognitions. Administered at baseline, post-treatment (week 12), and 6-month follow-up.
Change in WHOQOL-BREF global score | Baseline, Week 12 (post-treatment), 6-month follow-up
  26-item quality of life measure (scores 26-130). Higher scores indicate better QoL. Assessed at baseline, post-treatment, and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jiang Yingjie, PhD, Principal Investigator — Northeast Normal University, China
Locations (2):
- Pakistan (2):
  - IOMH Institute of Mental Health, Islamabad, Punjab Province
  - Subhan Medical Centre Trust, Islamabad, Punjab Province

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared publicly due to confidentiality and privacy concerns, as the data contains sensitive patient information. Additionally, institutional policies and legal restrictions prohibit the unrestricted distribution of raw data. Aggregate results will be made available in published manuscripts to ensure transparency

REFERENCES:
- [Background] Moritz S, Jelinek L, Hauschildt M, Naber D. How to treat the untreated: effectiveness of a self-help metacognitive training program (myMCT) for obsessive-compulsive disorder. Dialogues Clin Neurosci. 2010;12(2):209-20. doi: 10.31887/DCNS.2010.12.2/smoritz. PMID 20623925
- [Background] Philipp R, Kriston L, Lanio J, Kuhne F, Harter M, Moritz S, Meister R. Effectiveness of metacognitive interventions for mental disorders in adults-A systematic review and meta-analysis (METACOG). Clin Psychol Psychother. 2019 Mar;26(2):227-240. doi: 10.1002/cpp.2345. Epub 2018 Dec 16. PMID 30456821
- See also: Official publication of the myMCT manual used in this trial' — https://doi.org/10.1016/j.jocrd.2016.04.010